CLINICAL TRIAL: NCT03989297
Title: Expression and Clinical Significance of PD-L1 and BRAF Expression in Nasopharyngeal Carcinoma
Brief Title: PD-L1 and BRAF Expression in Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Kiang Wu Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KWH201701
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; programmed death-ligand 1; prognosis
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NPC patients: Consecutive patients who were pathologically diagnosed with NPC and for whom fresh-frozen tissue samples were available were included.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Consecutive patients who were pathologically diagnosed with NPC and treated with radiation at the Kiang Wu Hospital.

SUMMARY:
The prognostic value of programmed death-ligand 1 (PD-L1) and BRAF expression in nasopharyngeal carcinoma (NPC) is not well-defined. In this study the investigators investigated alterations in PD-L1, BRAF and EGFR by using immunohistochemistry analysis in a cohort of consecutively enrolled NPC patients.

DETAILED DESCRIPTION:
NPC is a common type cancer in Macau and Southern China. The role of PD-L1 in NPC remains controversial. There many reasons behind these inconsistent findings. We used the SP263 antibody with the standard cut off value of 1% and 5%, which is frequently used for lung cancer and other cancer types. We also plan to include over 150 patients, which will be the largest study in NPC. This will help us to gain insights in NPC.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Locally advanced (stage IIIB) or metastatic (stage IV) NPC
* Fresh-frozen tissue samples were available were included
* After treatment with curative surgery or radiotherapy in Macau
* With follow up data were available

Exclusion Criteria:

• Enrolment in studies that prohibit any participation in this observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who were pathologically diagnosed with NPC between 2006 and December 2010 at the Kiang Wu Hospital (Macau, SAR China) and for whom fresh-frozen tissue samples were available were included.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Response rate | Followed up with 12 months after last patient in
  Efficacy after radiation

SECONDARY OUTCOMES:
Survival rate | Followed up with 12 months after last patient in
  Survival in PD-L1 positive and negative group

CONTACTS AND LOCATIONS:
Overall Officials: Yabing Cao, MD; PhD, Principal Investigator — Kiang Wu Hospital, Department of Oncology
Locations (1):
- Kiang Wu Hospital, Macao, China

REFERENCES:
- [Derived] Cao Y, Chan KI, Xiao G, Chen Y, Qiu X, Hao H, Mak SC, Lin T. Expression and clinical significance of PD-L1 and BRAF expression in nasopharyngeal carcinoma. BMC Cancer. 2019 Oct 29;19(1):1022. doi: 10.1186/s12885-019-6276-y. PMID 31664962